CLINICAL TRIAL: NCT06953882
Title: SELECT: A Phase II Adjuvant Trial Evaluating the Impact of Omitting Chemotherapy Based on Patient's Selection for Moderate to High-Anatomical Risk, Low-Genomic Risk, ER-Positive, HER2- Negative Breast Cancer With a Combination Regimen of Ribociclib and Optimized Endocrine Therapy
Brief Title: Impact of Omitting Chemo Based on Patient's Selection for ER-Positive, HER2-Negative Breast Cancer With Ribociclib and Endocrine Therapy
Acronym: SELECT
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: Novartis (Industry); Breast Cancer Research Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2000038734; BCRF-23-184 (Other Grant/Funding Number: The Breast Cancer Research Foundation Inc.)
Record Dates: First submitted 2025-04-01; First posted 2025-05-01 (Actual); Last update posted 2025-07-14 (Actual); Status verified 2025-07

CONDITIONS: HER2 Negative Breast Cancer
Keywords: premenopausal women T1-3N1-2; postmenopausal women T3N1; postmenopausal women T3N2; ER-positive
MeSH Terms: interventions — ribociclib; Letrozole; Anastrozole; Goserelin; Chemotherapy, Adjuvant

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Ribociclib + Optimized Endocrine Therapy (Experimental): Combination of ribociclib and optimized endocrine therapy
  Interventions: Drug: Ribociclib 400mg; Drug: Letrozole 2.5mg; Drug: Anastrazole 1mg; Drug: Goserelin 3.6 MG
- Adjuvant Chemotherapy + Ribociclib & Optimized Endocrine Therapy (Experimental): Adjuvant chemotherapy followed by a combination of ribociclib and optimized endocrine therapy
  Interventions: Drug: Ribociclib 400mg; Drug: Letrozole 2.5mg; Drug: Anastrazole 1mg; Drug: Goserelin 3.6 MG; Radiation: Adjuvant chemotherapy

INTERVENTIONS:
Drug: Ribociclib 400mg — 400 mg (2 x 200 mg tablets by mouth) once daily on days 1 to 21 of a 28-day cycle, followed by seven days off ribociclib (Days 22 to 28).
Drug: Letrozole 2.5mg — Letrozole will be administered as an endocrine therapy. The regimen will differ depending on the demographic of the patient. For postmenopausal women: Letrozole 2.5 mg by mouth daily continuously. For men or premenopausal women: Letrozole 2.5 mg by mouth daily continuously.
Drug: Anastrazole 1mg — For postmenopausal women: Letrozole 2.5 mg by mouth daily continuously or anastrozole 1 mg by mouth daily continuously. For men or premenopausal women: Letrozole 2.5 mg by mouth daily continuously or anastrozole 1 mg by mouth daily continuously.
Drug: Goserelin 3.6 MG — For men or premenopausal women: Letrozole 2.5 mg by mouth daily continuously or anastrozole 1 mg by mouth daily continuously, concurrently with goserelin 3.6 mg monthly injection.
Radiation: Adjuvant chemotherapy — Adjuvant chemotherapy dose modifications in Arm 2 will be per institutional guidelines and investigator discretion.
  Arms: Adjuvant Chemotherapy + Ribociclib & Optimized Endocrine Therapy

SUMMARY:
This is a Phase II Trial to assess the impact of omitting adjuvant chemotherapy based on patient's selection on treatment persistence of CDK4/6 inhibitor, ribociclib (Kisqali), in a well-defined subgroup of patients with resected estrogen receptor (ER)-positive, HER2-negative, lymph node-positive breast cancer, but whose tumor profiling indicates a less aggressive biological nature (OncotypeDx 21-gene recurrence score RS 0-25).

DETAILED DESCRIPTION:
Most patients with ER-positive, HER2-negative, node-positive breast cancer are treated with curative intent, which typically involves some combination of surgery, radiation, endocrine therapy (ET) and often chemotherapy. The recent integration of CDK 4/6 inhibitors into adjuvant ET has complicated treatment decision-making for this subtype of breast cancer. These agents have demonstrated substantial benefits in reducing recurrence risk when combined with ET, prompting a reassessment of the role and necessity of chemotherapy in certain patient populations. However, it remains unclear to what extent prior exposure to a course of adjuvant chemotherapy impacts treatment persistence of CDK 4/6 inhibition. In the NATALEE and monarchE trials, approximately 90% of participants received prior chemotherapy, yet 28 - 36% participants discontinued the CDK 4/6 inhibitors prematurely. These findings underscore the significant barrier in maintaining long-term persistence to CDK 4/6 inhibitor therapy and emphasize the need to develop and implement strategies for optimizing treatment regimens to minimize discontinuation rates, especially in patients for whom the benefit of chemotherapy is uncertain.

This is a Phase II, two-arm, single center, patient preference clinical trial designed to evaluate the impact of omitting adjuvant chemotherapy on ribociclib treatment persistence in moderate to high-anatomical risk, low-genomic risk (Oncotype DX Recurrence Score, RS ≤ 25), ER-positive, HER2-negative breast cancer participants treated with a combination regimen of ribociclib and optimized endocrine therapy. Eligible participants aged ≥18 years, ECOG PS of 0 to 1, with anatomic stage II/III ER-positive (≥10%), HER2-negative breast cancer (men or premenopausal women with T1-3N1-2 or postmenopausal women with T3N1 or T1-3N2) and RS 0-25 will be included. Participants will have the option to decide whether to include adjuvant chemotherapy in their treatment plan. Arm 1 will receive the combination of ribociclib and optimized ET. Arm 2 will be treated with adjuvant chemotherapy followed by a combination of ribociclib and optimized ET. Optimized ET includes an oral aromatase inhibitor (letrozole or anastrozole) for all participants, with the addition of a GnRH agonist (goserelin) to achieve gonadal suppression in all men and premenopausal women. Key exclusion criteria are distant metastases, T4, N3, neoadjuvant chemotherapy and clinically significant uncontrolled heart disease at screening. The primary objective is to evaluate 1-year discontinuation rate of ribociclib in each arm. Secondary endpoints include 3-year invasive disease-free survival, factors impacting treatment decision, quality of life, decisional regret, and fear of recurrence. Estimated enrollment is 140 participants (70 each arm) to ensure investigators can estimate one-year discontinuation rate with a reasonable level of precision.

ELIGIBILITY:
Inclusion Criteria:

1. Female or male age ≥ 18 years old and have the ability to understand and the willingness to sign a written informed consent document.
2. Participants may have ipsilateral or contralateral synchronous breast cancer if the highest stage tumor meets entry criteria, and the other sites of disease would not require chemotherapy or HER2-directed therapy.
3. Participants may have multicentric or multifocal breast cancer if the highest stage tumor meets entry criteria, and the other sites of disease would not require chemotherapy or HER2-directed therapy.
4. Participants underwent a total mastectomy, skin-sparing mastectomy, nipple-sparing mastectomy, or a lumpectomy.
5. For participants who undergo a lumpectomy, the margins of the resected specimen or re-excision must be histologically free of invasive tumor and DCIS with no ink on tumor as determined by the local pathologist. If pathologic examination demonstrates tumor at the line of resection, additional excisions may be performed to obtain clear margins.

   a. Participants with margins positive for LCIS are eligible without additional resection.
6. For participants who undergo mastectomy, the margins must be free of residual gross tumor.

   a. Participants with microscopic positive margins are eligible if post mastectomy RT of the chest wall will be administered.
7. Participants must have undergone axillary staging with sentinel node biopsy (SNB), targeted axillary dissection (TAD), or axillary lymph node dissection (ALND).
8. The following staging criteria must be met postoperatively according to AJCC 8th edition criteria: Men or premenopausal women with T1-3N1-2. Postmenopausal women with T3N1 or T1-3N2 diseases.
9. The tumor must be ER-positive (≥ 10%), HER2-negative, by current ASCO/CAP guidelines based on testing results. HER2-negative breast cancer is defined as a negative in situ hybridization test or an immunohistochemistry (IHC) status of 0 or 1+. If IHC is 2+, a negative in situ hybridization (FISH, CISH, or SISH) test is required to confirm the participant's HER2-negative status (based on the most recently analyzed tissue sample tested by a local laboratory).
10. Oncotype Dx Recurrence Score must be 0 - 25.
11. Participants with known menopausal status at the time of screen.

    a. Postmenopausal status is defined as: i. Participant underwent bilateral oophorectomy, or ii. Age ≥ 60 years, or Age < 60 years and amenorrhea for 12 or more months (in the absence of chemotherapy, tamoxifen, toremifene or ovarian suppression) and Folliclestimulating hormone (FSH) and plasma estradiol are in the postmenopausal ranges per local normal ranges. Note: All women who do not meet the criteria for postmenopausal status are considered premenopausal for the purpose of this trial.
12. The interval between the last surgery for breast cancer (including re-excision of margins) and screening must be no more than 16 weeks.
13. HIV-infected participants with undetectable viral load within 6 months and in long term anti-retroviral therapy that would not have a significant drug-drug interaction with ribociclib are eligible for this trial.
14. Radiation therapy should be used according to standard guidelines.
15. Participants must have an ECOG performance status of 0 to 1 within 28 days prior to initiation of the study treatment.
16. Participant is able to swallow oral medications.
17. Participants must have adequate organ and marrow function as defined below. All laboratory values must be obtained within 14 days prior to screening.

    1. Absolute neutrophil count (ANC) ≥ 1.5 × 109/L.
    2. Platelets ≥ 100 × 109/L.
    3. Hemoglobin ≥ 9.0 g/dL.
    4. Estimated glomerular filtration rate (eGFR) ≥ 30 mL/min/1.73m2 according to the Modification of Diet in Renal Disease (MDRD) formula.
    5. Alanine transaminase (ALT) < 2.5 × Upper Limit Normal (ULN).
    6. Aspartate transaminase (AST) < 2.5 × ULN.
    7. Total serum bilirubin < ULN; or total bilirubin ≤ 3.0 × ULN or direct bilirubin ≤ 1.5 × ULN in patients with well documented Gilbert's Syndrome.
    8. International normalized ratio (INR) ≤ 1.5 (unless the patient is receiving anticoagulants, and the INR is within the therapeutic range of intended use for that anticoagulant within 7 days prior to enrollment).
    9. Patient must have the following laboratory values within normal limits or corrected to within normal limits with supplements (the local laboratory value should be documented within normal limits after the correction) before enrollment:

       * Potassium.
       * Magnesium.
       * Total Calcium (corrected for serum albumin).
18. Standard 12-lead ECG values assessed as: QTcF interval (using Fridericia's correction) at screening < 450 msec. Resting heart rate 50-90 beats per minute (determined from the ECG).
19. Participant must be willing and able to comply with scheduled visits, treatment plans, laboratory tests, and other trial procedures.
20. Participants must adhere to the following reproductive and contraceptive requirements while on study treatment and for the specified duration after the last dose of the treatment drugs.

    a. General requirements: i. Participants must not be pregnant or breastfeeding. ii. Participants must not donate or freeze eggs for future use related to assisted reproduction during the course of this study or within three months after receiving the last dose of the study treatment. b. For participants of childbearing potential: i. A participant of childbearing potential is defined as an individual who is premenopausal and capable of becoming pregnant. This includes individuals using contraception, those who are sexually inactive, and those with partners who have undergone a vasectomy. A participant is considered of childbearing potential if they have reached menarche, have not yet met the criteria for postmenopause (defined as more than 12 consecutive months of amenorrhea without any other medical cause), and have not undergone surgical sterilization (such as hysterectomy or oophorectomy).

    ii. A negative highly sensitive serum pregnancy test (for β-hCG) must be obtained within two weeks of starting the treatment drug administration.

    iii. Participants must practice at least one highly effective method of contraception.

    c. Highly effective methods of contraception include, but are not limited to: i. Total abstinence (no sexual relations), when this is in line with the participant's preferred and usual lifestyle. Periodic abstinence like calendar, ovulation, symptothermal, post-ovulation methods, and withdrawal are not acceptable methods of contraception.

    ii. Total hysterectomy (surgical removal of the uterus and cervix) or tubal ligation (participant's "tubes tied") at least six weeks before taking study treatment. iii. Participant's male partner has already been sterilized with the appropriate documentation. The sterilized male partner should be the sole partner.

    iv. Placement of an intrauterine device (IUD) v. The use of oral (estrogen and progesterone), injected or implanted hormonal methods of contraception or intrauterine system (IUS) or any other form of hormonal contraception (e.g., hormone vaginal ring, hormonal-based IUD or transdermal hormone contraception) is not allowed in this study.
21. Participant has no contraindication for the adjuvant ET in the trial and is planned to be treated with ET for five years or more.

Exclusion Criteria:

1. Definitive clinical or radiologic evidence of distant metastases of breast cancer beyond regional lymph nodes (stage IV according to AJCC 8th edition) and/or evidence of recurrence after curative surgery.
2. T4 tumors, including inflammatory breast cancer.
3. N3 tumors.
4. Participants that have received neoadjuvant chemotherapy or biotherapy.
5. Participant has received prior treatment with tamoxifen, raloxifene or AIs for reduction in risk ("chemoprevention") of breast cancer and/or treatment for osteoporosis within the last two years prior to randomization. Participant is concurrently using hormone replacement therapy.
6. Participants with a known hypersensitivity to any of the excipients of ribociclib and/or ET (e.g. rare hereditary problems of galactose intolerance, the Lapp lactase deficiency, glucose-galactose malabsorption, and soy allergy).
7. History of ipsilateral or contralateral invasive breast cancer: Participants with synchronous and/or previous ductal carcinoma in situ (DCIS) or lobular carcinoma in situ (LCIS) are eligible. If prior ipsilateral DCIS was treated with lumpectomy and radiation therapy, a mastectomy must have been performed for the current cancer.
8. Participant has received any CDK4/6 inhibitor.
9. Participant has a concurrent invasive malignancy or a prior invasive malignancy whose treatment was completed within two years before randomization. Note: Participants with adequately treated basal or squamous cell skin carcinoma or curatively resected cervical cancer in situ are eligible.
10. Participant has known active hepatitis B virus (HBV) or hepatitis C virus (HCV) infection (testing is not mandatory, unless required by local regulation).
11. Life expectancy of <10 years due to co-morbid conditions in the opinion of the treating investigator.
12. Non-epithelial breast malignancies such as sarcoma or lymphoma.
13. Hormonally based contraceptive measures must be discontinued prior to registration (including progestin/progesterone IUDs).
14. Pregnancy or lactating women or women who plan to become pregnant or breast-feed during the trial.

    a. Note: Pregnancy testing according to institutional standards for women of childbearing potential must be performed at screening.
15. Clinically significant, uncontrolled heart disease and/or cardiac repolarization abnormality, including any of the following:

    1. History of documented myocardial infarction (MI), angina pectoris, symptomatic pericarditis, or coronary artery bypass graft within six months prior to screening
    2. Documented cardiomyopathy
    3. Left Ventricular Ejection Fraction (LVEF) < 50% as determined by Multiple Gated acquisition (MUGA) scan or echocardiogram (ECHO) within six months prior to screening.
    4. Long QT syndrome or family history of idiopathic sudden death or congenital long QT syndrome, or any of the following:

    i. Risk factors for Torsades de Pointes (TdP) including uncorrected hypokalemia or hypomagnesemia, history of cardiac failure, or history of clinically significant/symptomatic bradycardia ii. Concomitant medication(s) with a known risk to prolong the QT interval and/or known to cause TdP that cannot be discontinued or replaced by safe alternative medication (e.g. within five half-lives or seven days prior to starting trial treatment) iii. Inability to determine the QTcF interval e. Clinically significant cardiac arrhythmias (e.g. ventricular tachycardia), complete left bundle branch block, high-grade Atrioventricular (AV) block (e.g.

    bifascicular block, Mobitz type II- and third-degree AV block) f. Uncontrolled arterial hypertension with systolic blood pressure > 160 mmHg.
16. Participant is currently receiving any of the following substances within 7 days before registration:

    1. Concomitant medications, herbal supplements, and/or fruits (e.g. grapefruit, pummelos, starfruit, Seville oranges) and their juices that are known as strong inhibitors or inducers of CYP3A4/5.
    2. Medications that have a narrow therapeutic window and are predominantly metabolized through CYP3A4/5.
17. Participant is currently receiving or has received systemic corticosteroids ≤ 2 weeks prior to starting trial treatment or has not fully recovered from side effects of such treatment.

    Note: The following uses of corticosteroids are permitted: a short duration (<5 days) of systemic corticosteroids, any duration of topical applications (e.g. for rash), inhaled sprays (e.g. for obstructive airways diseases), eye drops or local injections (e.g. intraarticular).
18. Participant has impairment of GI function or GI disease that may significantly alter the absorption of the oral trial treatments (e.g. uncontrolled ulcerative diseases, uncontrolled nausea, vomiting or diarrhea, malabsorption syndrome, or small bowel resection).
19. Participant has any other concurrent severe and/or uncontrolled medical condition that would, in the principal investigator's judgment, cause unacceptable safety risks, contraindicate patient participation in the clinical trial or compromise compliance with the protocol (e.g. chronic pancreatitis, chronic active hepatitis, liver cirrhosis or any other significant liver disease, active untreated or uncontrolled fungal, bacterial or viral infections, active infection requiring systemic anti-bacterial therapy, etc.) or limit life expectancy to ≤5 years.
20. Participation in other studies involving investigational drug(s) within 30 days prior to registration or within 5 half-lives of the investigational drug(s) (whichever is longer), or participation in any other type of medical research judged not to be scientifically or medically compatible with this trial. If the participant is enrolled or planned to be enrolled in another study that does not involve an investigational drug, the agreement of the Sponsor-Investigator is required to establish eligibility.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2025-07-09 (Actual); Primary Completion 2030-09 (Estimated); Study Completion 2030-09 (Estimated)

PRIMARY OUTCOMES:
Discontinuation rate of ribociclib in patients with resected moderate to high-anatomical risk, low-genomic risk, ER-positive, HER2-negative breast cancer | Within one year of treatment
  Discontinuation rate of ribociclib in participants with resected moderate to high-anatomical risk (men or premenopausal women T1-3N1-2, and postmenopausal women T3N1 or T1-3N2), low-genomic risk (RS≤ 25), ER-positive, HER2-negative breast cancer who choose to forgo or include adjuvant chemotherapy in their treatment regimen. One-year treatment discontinuation is defined as treatment discontinuation within one year for any reason (e.g., adverse events, disease recurrence, patient/investigator decision, lost to follow up, etc).

SECONDARY OUTCOMES:
Invasive disease-free survival in patients with resected moderate to high-anatomical risk, low-genomic risk, ER-positive, HER2-negative breast cancer | Defined as the time from initiation of treatment to three years post-survival
  iDFS is defined as the time from initiation of treatment to the first diagnosis of local invasive recurrence following mastectomy, local invasive recurrence in the ipsilateral breast following lumpectomy, regional recurrence, distant recurrence, contralateral invasive breast cancer, second non-breast primary cancer (excluding squamous or basal cell carcinoma of the skin), or death from any cause prior to recurrence or second primary cancer using STEEP criteria as assessed by investigator. iDFS using STEEP criteria, assessed separately in the participants who select to omit adjuvant chemotherapy (arm 1) and those who include adjuvant chemotherapy in their treatment regimen (arm 2).
Change from Baseline in Severity of Symptoms in patients with resected moderate to high-anatomical risk, low-genomic risk, ER-positive, HER2-negative breast cancer | At baseline, every three months during the first year and every six months during years 2 and 3
  This seeks to assess the change from baseline in the severity of symptoms. This will be measured using the Functional Assessment of Cancer Therapy-General (FACT-G) GP5. FACT-G GP5 will be scored from scale of 0-4; with 0 indicating "not at all" and 4 indicating "very much". The objective is to describe patient-reported outcomes (PRO) for these measures in participants in arm 1 and arm 2.
Change from Baseline in Physical Functioning and Global Health Status/Quality of Life in patients with resected moderate to high-anatomical risk, low-genomic risk, ER-positive, HER2-negative breast cancer | At baseline, every three months during the first year and every six months during years 2 and 3
  This seeks to evaluate the change from baseline in the physical functioning sub-scale score and global health status/Quality of Life scale score of participants. This will be measured using the European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire Core 30 (EORTC QLQ-C30). This questionnaire is scored from 1 to 4; with 1 indicating 'not at all' and 4 indicating 'very much'. The objective is to describe patient-reported outcomes related to health-related quality-of-life in participants in arm 1 and arm 2.
Factors Impacting Decision Making in Adjuvant Treatment Decisions in patients with resected moderate to high-anatomical risk, low-genomic risk, ER-positive, HER2-negative breast cancer | At baseline
  This seeks to to identify and understand the factors that impact participants' decision-making processes, as assessed by a modified version of the Control Preferences Scale. This tool uses a card-sorting method, where participants are asked to rank five cards with different decision-making roles. It is then scored by the participant's preference order over the five cards. The objective is to explore the factors influencing the decision to include or omit adjuvant treatment among participants in arm 1 and arm 2. This assessment will help in understanding the preferences and considerations of patients regarding their treatment plans.
Changes in fear of cancer recurrence in patients with resected moderate to high-anatomical risk, low-genomic risk, ER-positive, HER2-negative breast cancer | At baseline, six months, and one year
  This seeks to assess the changes in fear of cancer recurrence among participants, measured using the Fear of Cancer Recurrence-7 (FCR-7) scale. The first six items on the scale are scored on a 5-point scale, with 1 indicating "not at all" and 5 indicating "all the time". The seventh item assesses the extent to which Fear of Cancer Recurrence interferes with thoughts and activities on a 10 point scale, where 0 indicates "not at all" and 10 indicates "a great deal". The sale is then totaled; a score of less greater than 4 on items 1-6 or greater than 7 on item 7 suggests a significant level of fear of cancer recurrence. This evaluation aims to provide insights into the emotional and psychological impact of cancer treatment decisions.
Change from Baseline in Anxiety/Depression in patients with resected moderate to high-anatomical risk, low-genomic risk, ER-positive, HER2-negative breast cancer | At baseline, every three months during the first year and every six months during years 2 and 3
  This seeks to assess the change from baseline in anxiety and depression of participants. This will be measured using the Patient Health Questionnaire-9 (PHQ-9). PHQ-9 will be scored from 0 to 3, with 0 indicating 'not at all' and 3 indicating 'nearly every day'. The scores will then be tallied, with scores ranging from 0-27, where higher scores will indicate greater depression severity. The objective is to describe patient-reported outcomes (PRO) for these measures in participants in arm 1 and arm 2.
Changes in decision regret in patients with resected moderate to high-anatomical risk, low-genomic risk, ER-positive, HER2-negative breast cancer | At baseline, six months, and one year
  This seeks to assess the changes in decision regret among participants, measured using the Decision Regret Scale. This scale is scored from 1 to 5, where 1 indicates "strongly agree" and 5 indicates "strongly disagree". This evaluation aims to provide insights into the emotional and psychological impact of cancer treatment decisions
Change from Baseline in Severity of Symptoms in patients with resected moderate to high-anatomical risk, low-genomic risk, ER-positive, HER2-negative breast cancer | At baseline, every three months during the first year and every six months during years 2 and 3
  This seeks to assess the change from baseline in the severity of symptoms. This will be measured using the Common Terminology Criteria for Adverse Events-Patient Reported Outcome (CTCAE-PRO). CTCAE-PRO will be scored from "none/not at all" to "very severe/severe". The objective is to describe patient-reported outcomes (PRO) for these measures in participants in arm 1 and arm 2.

CONTACTS AND LOCATIONS:
Overall Officials: Jing Du, Principal Investigator — Yale University
Locations (1):
- Yale University, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No